CLINICAL TRIAL: NCT02601079
Title: Endodrill vs. Conventional Biopsy. Diagnostics and Genetic Analysis in Tumors of the Distal Esophagus and Cardia
Brief Title: Endodrill vs. Conventional Biopsy. Diagnostics and Genetic Analysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed very low possibility for significant differences between the two instruments.
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Martin Jeremiasen, Consultant Surgeon, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Endodrill I
Record Dates: First submitted 2015-10-27; First posted 2015-11-10 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Neoplasm
Keywords: Biopsy; Diagnostics; Genetic analysis
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional biopsy (Active Comparator): 4 out of 8 biopsies taken with a conventional biopsy forceps from the tumor tissue in the distal esophagus and cardia. The biopsies will be taken in random order "blinded" for the person performing the examination. 1 additional biopsy will be taken from the tumor tissue in order to be evaluated for appropriateness of further genetic analysis. Both type of biopsies will be taken from the same patient. In total 10 biopsies per patient.
  Interventions: Device: Conventional Biopsy forceps
- Endodrill biopsy (Active Comparator): 4 out of 8 biopsies taken with the Endodrill instrument from the tumor tissue in the distal esophagus and cardia. The biopsies will be taken in random order "blinded" for the person performing the examination. 1 additional biopsy will be taken from the tumor tissue in order to be evaluated for appropriateness of further genetic analysis. Both type of biopsies will be taken from the same patient. In total 10 biopsies per patient.
  Interventions: Device: Endodrill Biopsy

INTERVENTIONS:
Device: Endodrill Biopsy — Testing a new device for taking tissue biopsies in the GI tract. The investigators will use the Endodrill instrument in order to sample high quality biopsies from tumor tissue in the distal esophagus and cardia. The investigators will also investigate to what extent the Endodrill instrument can generate biopsies with the correct diagnosis and also evaluate the possibility for genetic studies of the harvested tumor tissue.
  Arms: Endodrill biopsy
Device: Conventional Biopsy forceps — Using a conventional biopsy forceps for taking tissue biopsies in the GI tract. The investigators will use conventional biopsy forceps in order to sample high quality biopsies from tumor tissue in the distal esophagus and cardia. The investigators will also investigate to what extent the conventional biopsy forceps can generate biopsies with the correct diagnosis and also evaluate the possibility for genetic studies of the harvested tumor tissue.
  Arms: Conventional biopsy

SUMMARY:
Endodrill is a new instrument for biopsy sampling in the GI-channel. The purposes of this study are as follows:

* Compare the Endodrill instrument with conventional biopsy forceps in terms of ability to establish the correct diagnosis based on collected biopsies of tumors in the upper GI tract.
* Based on the quality of the collected tissue samples we want to evaluate which instrument generates the most useful material for genetic studies of the tumor.

DETAILED DESCRIPTION:
Endodrill is a newly constructed biopsy tool for flexible endoscopic use. It uses a drilling motion within a casing to harvest solid biopsies from tissue through the biopsy channel of a conventional flexible endoscope. It was originally designed for sampling of tissue from submucosal lesions. The investigators´ first study of the instrument is now finished. Endodrill is safe to use and generates more submucosal tissue compared to biopsies with a conventional biopsy forceps.

In this study the investigators want to compare the Endodrill instrument´s ability to obtain representative tissue samples from tumors in the distal esophagus and cardia with a conventional biopsy forceps. In addition the investigators want to compare the tissue samples in terms of weight, quality, artefacts and whether either instrument is more suited for collecting tissue for genetic analysis. Such analysis will be conducted with Next-Generation Sequensing (NGS) of the whole exome, Whole Exome Sequensing (WES). In the event of positive results from these analysis the investigators will also conduct RNA-sequencing of the tumor tissue in order to start pre-operative mapping of genetic abnormalities.

20 patients will be enrolled for this study. For each patient the investigators will collect 10 biopsies, 5 biopsies each with conventional biopsy and the Endodrill instrument respectively. The order will be randomized for each patient. For each specific biopsy the investigator will choose a particular site on the suspected tumor tissue without knowing which instrument that will be used for the biopsy. This procedure will be repeated for all 10 biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with adenocarcinoma of the distal esophagus/cardia or stomach capable of stating a formal consent to participate in the study.

Exclusion Criteria:

* Mental illness
* Extreme co-morbidity (ASA >3)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Highest proportion (number) of representative biopsies for diagnostic purposes from the tumor tissue. | 12 months

SECONDARY OUTCOMES:
Number of genetic point mutations in tissue harvested from esophageal neoplasms prior to neoadjuvant oncological treatment. | 12 months
Number of fusion genes in tissue harvested from esophageal neoplasms prior to neoadjuvant oncological treatment. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Johansson, SrConsultant, Principal Investigator — Region Skåne
Locations (1):
- University Hospital of Lund, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No